CLINICAL TRIAL: NCT00532662
Title: Intravenous Versus Caudal Supplementation of Ketamine for Postoperative Pain Control in Children,A Double-blind Controlled Clinical Trial.
Brief Title: Postoperative Analgesia by Epidural vs IV Ketamine Concurrent With Caudal Anesthesia in Pediatric Orthopedic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: HamidReza Amiri/Assistant professor, TehranUMS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 86-02-78-56790
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Analgesia
Keywords: Epidural; Intravenous; Ketamine; Analgesia; Caudal; Pediatric; Regional; Local Anesthetics
MeSH Terms: conditions — Agnosia | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): epidural s(+)-ketamine for supplementation of caudal anesthesia
  Interventions: Drug: S(+)-ketamine
- 2 (Active Comparator): intravenous ketamine for supplementation of caudal anesthesia
  Interventions: Drug: S(+)-ketamine

INTERVENTIONS:
Drug: S(+)-ketamine — epidural or intravenous 1 mg kg-1 once concurrent with caudal anesthesia

SUMMARY:
Preemptive analgesia can improve postoperative pain management. Ketamine may prevent central sensitization during surgery and result in preemptive analgesia. The purpose of this study is to examine the effectiveness of ketamine as a preemptive analgesic as previous studies have shown the involvement of N-methyl-D-Aspartate (NMDA) receptor in neuroplasticity.

DETAILED DESCRIPTION:
After receiving consent inform from parents, 40 children scheduled for orthopedic surgeries will be randomized to one of two groups: epidural group and intravenous group, both will receive 1 mg kg-1 S(+)-ketamine. All patients will receive caudal block anesthesia with marcaine. Cardiovascular monitoring will be assessed during operation. Follow up will continue for 24 hours after caudal block. Duration of analgesia, first time of analgesic request and complications will be recorded by an orthopedic assistant that is blinded to study. Data will be analyzed statistically by Chi square, t test and nonparametric tests.

ELIGIBILITY:
Inclusion Criteria:

* Children aged < = 12 years
* Children scheduled for elective orthopedic surgery with caudal block
* ASA score < = 3

Exclusion Criteria:

* Contraindication for caudal block such as vertebral defect or infection at the site of block
* Disagreement of parents
* Patient's age > 12 years
* ASA score > = 4

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-06 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
pain score | 24 hours after anesthesia

SECONDARY OUTCOMES:
analgesic request | 24 hours after anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Espandar, MD, Study Chair — Imam Khomeini hospital- tehran university of medical sciences
Locations (2):
- Iran (2):
  - orthopedic ward of Imam Khomeini hospital, Tehran, Tehran Province
  - orthopedic surgery room- Imam Khomeini hospital, Tehran, Tehran Province